CLINICAL TRIAL: NCT00952679
Title: Computed Tomography (CT) Based Lymphatic Mapping and Localization of Sentinel Lymph Node in Breast Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Fudan University Cancer institue, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FCW001
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Breast Cancer
Keywords: The investigators evaluated the new method by comparing lymph nodes defined by CT and traditional ways.
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental arm (Experimental)
  Interventions: Device: Breast Lesion Localization Needles (interv)

INTERVENTIONS:
Device: Breast Lesion Localization Needles (interv) — needles to locate sln in CT monitor guided by CT

SUMMARY:
Breast cancer patients who diagnosed by core needle biopsy or excisional biopsy underwent CT scan to locate the sentinel lymph node (SLN) before SLN biopsy (SLNB) at the same day of surgery. When CT examination performed, those patients were in supine position, with the arms stretched upward but bent at the elbow with the hands at the side of the cranium which similar to the surgical position. After local anesthesia, 2mL of iopamidol was injected subcutaneously to the peritumoral and peri-areolar areas followed by gentle massage for about 1 minute. Contiguous 2-mm-thick CT images that included the breast and axilla were obtained prior to administration of the contrast agent. After 3D CT reconstruction, the SLN was identified as the most inferiorly visible nodule in the axilla connected to the lymphatic vessel on the CT imaging monitor. A professional intervention doctor punctured the defined lymph node guided by the CT monitor using the Breast Lesion Localization Needles (interv). The needle would stay in the patient's axilla until the surgery. All the lymph nodes including the CT defined one and which marked by methylene blue dye or 99mTc-sulfur colloid tracers were removed, which then would be tested by touch imprint cytology for the intraoperative diagnosis. Patients who had positive SLN would receive axillary dissection. The investigators evaluated the new method by comparing lymph nodes defined by CT and traditional ways.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients（T1-T2N0）
* Age 18-70
* Accept of SLNB
* Accept our protocol in the informed consent

Exclusion Criteria:

* LABC patients
* Age < 18
* History of epilepsy
* History of thyrotoxicosis
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-01 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | five years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital, Shanghai, Shanghai Municipality, China